CLINICAL TRIAL: NCT00918788
Title: Laser Spectroscopy of Breast Tissue Through a Needle Device
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE9107; P30CA043703 (NIH); CASE9107 (Other: Case Comprehensive Cancer Center); CASE-9107-CC482 (Other: Case Cancer IRB)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Immunohistochemistry; Microscopy; Biopsy, Needle; Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This laboratory study is looking at samples of breast tissue from women who have undergone breast biopsy or surgery.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: biologic sample preservation procedure — Ex vivo samples of normal and malignant breast tissue; biopsy specimens are then fixed in formalin and submitted for histopathologic studies
Other: immunohistochemistry staining method — The biopsy specimens are then fixed in formalin and submitted for histopathologic studies using standard light microscopy techniques (i.e., H&E staining and IHC). Additional histochemical, immunohistochemical, and fluorescent in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.
Other: light microscopy — The biopsy specimens are then fixed in formalin and submitted for histopathologic studies using standard light microscopy techniques (i.e., H&E staining and IHC).
Other: medical chart review — Medical records are reviewed to obtain information from the pathology report on patient demographics, pathological characteristics of the surgical specimen, and clinical indication for the surgical procedure.
Procedure: histopathologic examination — The biopsy specimens are then fixed in formalin and submitted for histopathologic studies using standard light microscopy techniques (i.e., H&E staining and IHC). Additional histochemical, immunohistochemical, and fluorescent in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.
Procedure: needle biopsy — Tissue spectra are measured using a portable clinical spectroscopy device with front- and side-viewing optical fiber probes that are inserted into the breast tissue through a hollow biopsy needle.
Procedure: spectroscopy — Optical spectra are acquired from ex vivo samples of normal and malignant breast tissue using diffuse reflectance, fluorescence, and Raman spectroscopy. Tissue spectra are measured using a portable clinical spectroscopy device with front- and side-viewing optical fiber probes that are inserted into the breast tissue through a hollow biopsy needle. After the probes are withdrawn through the needle, cutting biopsies are obtained and the tissue is marked at the site of the spectral measurements.

SUMMARY:
RATIONALE: Collecting and storing samples of breast tissue from patients who have undergone biopsy or surgery to test in the laboratory may help the study of cancer in the future.

PURPOSE: This laboratory study is looking at samples of breast tissue from women who have undergone breast biopsy or surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To prove that optical spectra collected by inserting an optical fiber probe into breast tissue through a biopsy needle can be of adequate quality to render a spectroscopic diagnosis.

OUTLINE: Optical spectra are acquired from ex vivo samples of normal and malignant breast tissue using diffuse reflectance, fluorescence, and Raman spectroscopy. Tissue spectra are measured using a portable clinical spectroscopy device with front- and side-viewing optical fiber probes that are inserted into the breast tissue through a hollow biopsy needle. After the probes are withdrawn through the needle, cutting biopsies are obtained and the tissue is marked at the site of the spectral measurements. The biopsy specimens are then fixed in formalin and submitted for histopathologic studies using standard light microscopy techniques (i.e., H&E staining and IHC). Additional histochemical, immunohistochemical, and fluorescent in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.

Medical records are reviewed to obtain information from the pathology report on patient demographics, pathological characteristics of the surgical specimen, and clinical indication for the surgical procedure.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Discarded normal and malignant breast tissue surgical specimens from women who have undergone excisional breast biopsy, lumpectomy, mastectomy, or breast-reduction surgery at the University Hospitals-Case Medical Center
* Hormone receptor status unknown

PATIENT CHARACTERISTICS:

* Menopausal status unknown

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Collection of optical spectra from normal and malignant breast tissue samples | at time of excisional breast biopsy, lumpectomy, mastectomy or breast reduction surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maryann Fitzmaurice, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States